CLINICAL TRIAL: NCT00357903
Title: Open-Label Extension Treatment With Tumor Necrosis Factor Receptor Fusion Protein (TNFR:Fc) for Participating Patients in Tumor Necrosis Factor Receptor Fusion Protein (TNFR:Fc) Clinical Trials
Brief Title: Open-Label Extension Treatment With Etanercept (TNFR:Fc) for Participating Patients in Etanercept (TNFR:Fc) Clinical Trials
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Immunex Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20021618; 16.0018
Record Dates: First submitted 2006-07-26; First posted 2006-07-28 (Estimated); Results first posted 2010-12-06 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis, Etanercept, Long-term Safety, Enbrel
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

ARMS (1):
- 1 (Other)
  Interventions: Biological: Etanercept

INTERVENTIONS:
Biological: Etanercept — Adult Rheumatoid Arthritis (RA) patients on etanercept (TNFR:Fc) with well controlled arthritic symptoms will continue on the etanercept (TNFR:Fc) dose administered in their original protocol of enrollment. All other adults will receive 50 mg per week as two 25 mg subcutaneous (SC) injections at separate sites, either on the same day or 3 or 4 days apart. Pediatric patients ages 4 to 17 years will receive a 0.8 mg/kg per week dose (up to a maximum of 50 mg per week).

SUMMARY:
This study was designed to provide all adult and pediatric arthritis patients (placebo and etanercept(TNFR:Fc) treated) who have participated in clinical trials with etanercept (TNFR:Fc) the opportunity to receive continued treatment with etanercept (TNFR:Fc). The primary objective of this study is to examine safety parameters.

ELIGIBILITY:
Inclusion Criteria:

* Previous enrollment in Immunex protocols
* No clinically significant adverse events thought to be due to etanercept (TNFR:Fc) during previous treatment.
* Negative serum pregnancy test not more than 14 days before the first dose of study drug in females of childbearing potential.
* No more than one NSAID at a dose not greater than the maximum recommended dose and stable for at least two weeks prior to administration of etanercept (TNFR:Fc). Exclusion Criteria: - Previous receipt of TNFR:Fc (p55), antibody to TNF, anti-CD4 antibody, or diphtheria IL-2 fusion protein.
* Receipt of investigational drugs or biologics (other than TNFR:Fc [p75]) within 1 month prior to the first dose of etanercept (TNFR:Fc) in this study.
* Receipt of DMARDs or methotrexate (except patients from 16.0014) within two weeks prior to the first dose of etanercept (TNFR:Fc) in this study.
* Receipt of cyclophosphamide within six months prior to the first dose of (etanercept (TNFR:Fc) in this study.
* Receipt of cyclosporin within two weeks prior to the first dose of etanercept (TNFR:Fc) in this study.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 639 (Actual)
Dates: Start 1997-04; Primary Completion 2008-12 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Fleischmann RM, Baumgartner SW, Tindall EA, Weaver AL, Moreland LW, Schiff MH, Martin RW, Spencer-Green GT. Response to etanercept (Enbrel) in elderly patients with rheumatoid arthritis: a retrospective analysis of clinical trial results. J Rheumatol. 2003 Apr;30(4):691-6. PMID 12672185
- [Background] Kremer JM, Weinblatt ME, Bankhurst AD, Bulpitt KJ, Fleischmann RM, Jackson CG, Atkins KM, Feng A, Burge DJ. Etanercept added to background methotrexate therapy in patients with rheumatoid arthritis: continued observations. Arthritis Rheum. 2003 Jun;48(6):1493-9. doi: 10.1002/art.11142. PMID 12794815
- [Background] Lovell DJ, Giannini EH, Reiff A, Jones OY, Schneider R, Olson JC, Stein LD, Gedalia A, Ilowite NT, Wallace CA, Lange M, Finck BK, Burge DJ; Pediatric Rheumatology Collaborative Study Group. Long-term efficacy and safety of etanercept in children with polyarticular-course juvenile rheumatoid arthritis: interim results from an ongoing multicenter, open-label, extended-treatment trial. Arthritis Rheum. 2003 Jan;48(1):218-26. doi: 10.1002/art.10710. PMID 12528122
- [Background] Lovell DJ, Reiff A, Ilowite NT, Wallace CA, Chon Y, Lin SL, Baumgartner SW, Giannini EH; Pediatric Rheumatology Collaborative Study Group. Safety and efficacy of up to eight years of continuous etanercept therapy in patients with juvenile rheumatoid arthritis. Arthritis Rheum. 2008 May;58(5):1496-504. doi: 10.1002/art.23427. PMID 18438876
- [Background] Lovell DJ, Reiff A, Jones OY, Schneider R, Nocton J, Stein LD, Gedalia A, Ilowite NT, Wallace CA, Whitmore JB, White B, Giannini EH; Pediatric Rheumatology Collaborative Study Group. Long-term safety and efficacy of etanercept in children with polyarticular-course juvenile rheumatoid arthritis. Arthritis Rheum. 2006 Jun;54(6):1987-94. doi: 10.1002/art.21885. PMID 16732547
- [Background] Moreland LW, Bucy RP, Weinblatt ME, Mohler KM, Spencer-Green GT, Chatham WW. Immune function in patients with rheumatoid arthritis treated with etanercept. Clin Immunol. 2002 Apr;103(1):13-21. doi: 10.1006/clim.2001.5183. PMID 11987981
- [Background] Moreland LW, Cohen SB, Baumgartner SW, Tindall EA, Bulpitt K, Martin R, Weinblatt M, Taborn J, Weaver A, Burge DJ, Schiff MH. Long-term safety and efficacy of etanercept in patients with rheumatoid arthritis. J Rheumatol. 2001 Jun;28(6):1238-44. PMID 11409115
- [Background] Moreland LW, Weinblatt ME, Keystone EC, Kremer JM, Martin RW, Schiff MH, Whitmore JB, White BW. Etanercept treatment in adults with established rheumatoid arthritis: 7 years of clinical experience. J Rheumatol. 2006 May;33(5):854-61. Epub 2006 Mar 15. PMID 16541481
- [Background] Stone JH, Uhlfelder ML, Hellmann DB, Crook S, Bedocs NM, Hoffman GS. Etanercept combined with conventional treatment in Wegener's granulomatosis: a six-month open-label trial to evaluate safety. Arthritis Rheum. 2001 May;44(5):1149-54. doi: 10.1002/1529-0131(200105)44:53.0.CO;2-F. PMID 11352248
- [Derived] Weinblatt ME, Bathon JM, Kremer JM, Fleischmann RM, Schiff MH, Martin RW, Baumgartner SW, Park GS, Mancini EL, Genovese MC. Safety and efficacy of etanercept beyond 10 years of therapy in North American patients with early and longstanding rheumatoid arthritis. Arthritis Care Res (Hoboken). 2011 Mar;63(3):373-82. doi: 10.1002/acr.20372. Epub 2010 Oct 18. PMID 20957659
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 31 July 1997 through 12 Oct 1999
Groups:
- Adult Participants: Adult participants with rheumatoid arthritis treated with a maximum etanercept dose of 50 mg administered subcutaneously once weekly
- Pediatric Participants: Pediatric participants with juvenile rheumatoid arthritis who received a maximum 50 mg dose of etanercept administered subcutaneously once weekly
Period: Overall Study
Arm/Group | Adult Participants | Pediatric Participants
Started | 581 | 58
Completed | 218 | 15
Not Completed | 363 | 43
Not completed — Adverse Event | 87 | 4
Not completed — Death | 33 | 0
Not completed — Lost to Follow-up | 23 | 4
Not completed — Physician Decision | 39 | 5
Not completed — Withdrawal by Subject | 57 | 7
Not completed — Completed month 12 only | 0 | 1
Not completed — Protocol issues | 14 | 3
Not completed — Response status | 61 | 9
Not completed — Other | 49 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pediatric Participants | Adult Participants | Total
Number analyzed (Participants) | 58 | 581 | 639
Age, Continuous [Mean (Standard Deviation); unit: Years] | 11.02 (3.80) | 52.87 (12.03) | 49.07 (16.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 465 | 504
  Male | 19 | 116 | 135
Race/Ethnicity, Customized [Number; unit: Participant]
  American Indian or Alaska Native | 1 | 4 | 5
  Asian | 1 | 10 | 11
  Black or African American | 4 | 18 | 22
  Hispanic or Latino | 9 | 25 | 34
  White or Caucasian | 43 | 522 | 565
  Other | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Total Exposure to Etanercept With Gaps
Description: Total participant exposure to etanercept (Enbrel) with gaps
Time Frame: Up to 10 years
Population: All participants who received at least one dose of etanercept
Measure: Number; unit: Participant-years
Arm/Group | Adult Participants | Pediatric Participants
Number analyzed (Participants) | 581 | 58
Participant-years | 4033.07 | 341.98

2. Secondary Outcome: Dosing Period
Description: Duration of etanercept dosing
Time Frame: Up to 10 years
Population: All participants who received at least one dose of etanercept
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Adult Participants | Pediatric Participants
Number analyzed (Participants) | 581 | 58
Days | 2535.4 (1433.77) | 2153.6 (1379.15)

3. Primary Outcome: Total Exposure Adjusted Rate of Malignancies
Description: Exposure-adjusted rate of malignancies, excluding nonmelanoma skin cancers, occurring on study within 30 days of the last dose of etanercept
Time Frame: Up to 10 years
Population: All participants who received at least one dose of etanercept
Measure: Number; unit: Malignancies per 100 participant-years
Arm/Group | Adult Participants | Pediatric Participants
Number analyzed (Participants) | 581 | 58
Malignancies per 100 participant-years | 1.41 | 0.00

4. Primary Outcome: Total Exposure Adjusted Rate of Deaths
Description: Rate of deaths within 30 days of the last dose of etanercept, adjusted for total exposure to etanercept
Time Frame: Up to 10 years
Population: All participants who received at least one dose of etanercept
Measure: Number; unit: Deaths per 100 participant-years
Arm/Group | Adult Participants | Pediatric Participants
Number analyzed (Participants) | 581 | 58
Deaths per 100 participant-years | 0.57 | 0.00

5. Primary Outcome: Total Exposure Adjusted Rate of Serious Infectious Events
Description: Exposure-adjusted rate of serious infectious events (associated with hospitalization or IV antibiotics) occurring on study within 30 days of the last dose of etanercept
Time Frame: Up to 10 years
Population: All participants who received at least one dose of etanercept
Measure: Number; unit: Events per 100 participant-years
Arm/Group | Adult Participants | Pediatric Participants
Number analyzed (Participants) | 581 | 58
Events per 100 participant-years | 5.18 | 3.22

6. Primary Outcome: Total Exposure Adjusted Rate of Lymphomas
Description: Rate of lymphomas occurring on study within 30 days of the last dose of etanercept, adjusted for total exposure to etanercept
Time Frame: Up to 10 years
Population: All participants who received at least one dose of etanercept
Measure: Number; unit: Lymphomas per 100 participant-years
Arm/Group | Adult Participants | Pediatric Participants
Number analyzed (Participants) | 581 | 58
Lymphomas per 100 participant-years | 0.15 | 0.00

7. Primary Outcome: Malignancy
Description: Occurrence of one or more malignancies on study within 30 days of the last dose of etanercept
Time Frame: Up to 10 years
Population: All participants who received at least one dose of etanercept
Measure: Number; unit: Participants
Arm/Group | Adult Participants | Pediatric Participants
Number analyzed (Participants) | 581 | 58
Participants | 48 | 0

8. Primary Outcome: Lymphoma
Description: Occurrence of one or more lymphomas on study within 30 days of the last dose of etanercept
Time Frame: Up to 10 years
Population: All participants who received at least one dose of etanercept
Measure: Number; unit: Participants
Arm/Group | Adult Participants | Pediatric Participants
Number analyzed (Participants) | 581 | 58
Participants | 6 | 0

9. Primary Outcome: Serious Infectious Event
Description: Occurrence of one or more serious infectious events within the participant on study within 30 days of the last dose of study medication. A serious infectious event is a serious adverse event that is infectious.
Time Frame: Up to 10 years
Population: All participants who received at least one dose of etanercept
Measure: Number; unit: Participants
Arm/Group | Adult Participants | Pediatric Participants
Number analyzed (Participants) | 581 | 58
Participants | 114 | 8

10. Primary Outcome: Death
Description: Occurrence of death on study within 30 days of the last dose of etanercept
Time Frame: Up to 10 years
Population: All participants who received at least one dose of etanercept
Measure: Number; unit: Participants
Arm/Group | Adult Participants | Pediatric Participants
Number analyzed (Participants) | 581 | 58
Participants | 23 | 0

11. Secondary Outcome: Tender Joint Count
Description: Number of tender joints, as assessed by the investigator using criteria based on pressure and joint manipulation
Time Frame: Month 12
Population: All participants who received at least one dose of etanercept and had available data
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Adult Participants | Pediatric Participants
Number analyzed (Participants) | 509 | 15
Joints | 9.55 (10.97) | 11.60 (10.61)

12. Secondary Outcome: Swollen Joint Count
Description: Number of swollen joints
Time Frame: Month 12
Population: All participants who received at least one dose of etanercept and had available data
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Adult Participants | Pediatric Participants
Number analyzed (Participants) | 510 | 28
Joints | 9.14 (8.83) | 11.93 (11.86)

13. Secondary Outcome: Health Assessment Questionnaire Disability Index
Description: Health Assessment Questionnaire Disability Index (HAQ DI). This index is a weighted average of 24 items, each scored 0 (no difficulty) to 3 (unable to function).
Time Frame: Month 12
Population: All participants who received at least one dose of etanercept and had available data
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Adult Participants
Number analyzed (Participants) | 485
Units on a scale | 0.96 (0.71)

14. Secondary Outcome: Childhood Health Assessment Questionnaire
Description: Childhood Health Assessment Questionnaire (CHAQ) disability index, having a range of 0 (no difficulty) to 3 (unable to do).
Time Frame: Month 12
Population: All participants who received at least one dose of etanercept and had available data
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pediatric Participants
Number analyzed (Participants) | 46
Units on a scale | 1.08 (0.95)

15. Secondary Outcome: C-Reactive Protein
Description: C-reactive protein at month 12
Time Frame: Month 12
Population: All participants who received at least one dose of etanercept and had available data
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Adult Participants | Pediatric Participants
Number analyzed (Participants) | 509 | 48
mg/dL | 1.37 (1.85) | 2.11 (3.82)

16. Secondary Outcome: ACR20 at Month 3 in Adults
Description: American College of Rheumatology (ACR) 20, defined as a 20% improvement in both tender and swollen joints (78 joints) and a 20% improvement in 3 of 5 items (including physician and patient global assessments), in adults
Time Frame: Baseline and month 3
Population: All participants who received at least one dose of etanercept and had available data at both baseline and month 3
Measure: Number; unit: Participants
Arm/Group | Adult Participants
Number analyzed (Participants) | 560
Participants | 372

17. Secondary Outcome: JRA DOI 30 at Month 3 in Juveniles
Description: Juvenile Rheumatoid Arthritis Definition of Improvement 30 (JRA DOI 30), defined as a 30% improvement from baseline in 3 of 6 items (including Childhood Health Assessment Questionnaire, disease severity, overall well-being, and erythrocyte sedimentation rate) and a worsening of >30% in at most one of the remaining items.
Time Frame: Baseline and month 3
Population: All participants who received at least one dose of etanercept and were evaluable for this endpoint at 3 months
Measure: Number; unit: Participants
Arm/Group | Pediatric Participants
Number analyzed (Participants) | 53
Participants | 46

18. Secondary Outcome: Standardized Incidence Rate for All SEER Cancers
Description: Standardized incidence rate for all cancers tracked by the National Cancer Institute's Surveillance Epidemiology and End Results (SEER) system.
Time Frame: up to 10 years
Population: All participants who received at least one dose of etanercept
Measure: Number; unit: Observed count / expected count
Arm/Group | Adult Participants | Pediatric Participants
Number analyzed (Participants) | 581 | 58
Observed count / expected count | 1.30 | 0.00
Statistical Analysis 1: Comparison: Pediatric Participants; Test type: Superiority or Other; Standardized incidence rate = 0.00, 95% CI [0.00 to 53.87]
Statistical Analysis 2: Comparison: Adult Participants; Test type: Superiority or Other; Standardized incidence rate = 1.30, 95% CI [0.97 to 1.71]

19. Primary Outcome: Total Exposure Adjusted Rate of Serious Adverse Events
Description: Rate of serious adverse events adjusted to total exposure to etanercept (events / exposure * 100)
Time Frame: Up to 10 years
Population: All participants who received at least one dose of etanercept
Measure: Number; unit: Events per 100 participant-years
Arm/Group | Adult Participants | Pediatric Participants
Number analyzed (Participants) | 581 | 58
Events per 100 participant-years | 20.95 | 12.87

ADVERSE EVENTS:
Time Frame: Up to 11.29 years
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Total Adults | Pediatric Subjects
Serious Adverse Events (participants affected / at risk) | 293/581 | 16/58
Other Adverse Events (participants affected / at risk) | 484/581 | 49/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total Adults (N=581) | Pediatric Subjects (N=58)
Anaemia (Blood and lymphatic system disorders) | 6 | 0
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0
Splenic infarction (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 3 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 7 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 5 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 13 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 12 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Cyanosis (Cardiac disorders) | 1 | 0
Diastolic dysfunction (Cardiac disorders) | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 20 | 0
Myocarditis (Cardiac disorders) | 2 | 0
Pericarditis (Cardiac disorders) | 2 | 0
Sick sinus syndrome (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 2 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal hernia obstructive (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Colitis (Gastrointestinal disorders) | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Diverticulum oesophageal (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 4 | 0
Gastroduodenitis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Large intestine perforation (Gastrointestinal disorders) | 2 | 0
Oesophageal rupture (Gastrointestinal disorders) | 2 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Rectal prolapse (Gastrointestinal disorders) | 1 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 2 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Adverse event (General disorders) | 1 | 0
Asthenia (General disorders) | 4 | 0
Chest discomfort (General disorders) | 2 | 0
Chest pain (General disorders) | 10 | 0
Condition aggravated (General disorders) | 25 | 3
Death (General disorders) | 4 | 0
Fatigue (General disorders) | 1 | 0
Impaired healing (General disorders) | 1 | 0
Necrosis (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 3 | 0
Oedema peripheral (General disorders) | 2 | 0
Pain (General disorders) | 3 | 0
Pyrexia (General disorders) | 4 | 1
Sudden death (General disorders) | 1 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 5 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 5 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatitis alcoholic (Hepatobiliary disorders) | 1 | 0
Perforation bile duct (Hepatobiliary disorders) | 1 | 0
Allergy to arthropod sting (Immune system disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1
Sarcoidosis (Immune system disorders) | 1 | 0
Abdominal infection (Infections and infestations) | 2 | 0
Abscess (Infections and infestations) | 1 | 0
Abscess intestinal (Infections and infestations) | 1 | 0
Abscess limb (Infections and infestations) | 3 | 0
Appendicitis (Infections and infestations) | 1 | 1
Arthritis bacterial (Infections and infestations) | 9 | 0
Arthritis infective (Infections and infestations) | 4 | 0
Atypical mycobacterial infection (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 4 | 0
Bronchopneumonia (Infections and infestations) | 3 | 0
Bursitis infective (Infections and infestations) | 4 | 0
Cellulitis (Infections and infestations) | 19 | 0
Cellulitis staphylococcal (Infections and infestations) | 1 | 0
Cellulitis streptococcal (Infections and infestations) | 2 | 0
Clostridium difficile colitis (Infections and infestations) | 2 | 0
Diarrhoea infectious (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 7 | 0
Enterocolitis infectious (Infections and infestations) | 3 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Fungal sepsis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 2 | 0
Graft infection (Infections and infestations) | 1 | 0
Hepatitis B (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 3 | 2
Incisional hernia gangrenous (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 6 | 0
Influenza (Infections and infestations) | 3 | 0
Kidney infection (Infections and infestations) | 2 | 0
Localised infection (Infections and infestations) | 2 | 0
Lung infection (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 1 | 0
Meningitis aseptic (Infections and infestations) | 1 | 1
Meningococcal sepsis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 3 | 0
Peritonitis bacterial (Infections and infestations) | 1 | 1
Pneumococcal sepsis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 36 | 0
Post procedural infection (Infections and infestations) | 3 | 1
Post procedural pneumonia (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 1
Proteus infection (Infections and infestations) | 1 | 0
Pseudomembranous colitis (Infections and infestations) | 2 | 0
Pyelonephritis (Infections and infestations) | 6 | 1
Sepsis (Infections and infestations) | 10 | 1
Sepsis syndrome (Infections and infestations) | 2 | 1
Septic shock (Infections and infestations) | 1 | 0
Shigella infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 2 | 0
Skin infection (Infections and infestations) | 14 | 2
Soft tissue infection (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 5 | 0
Staphylococcal skin infection (Infections and infestations) | 1 | 0
Streptococcal infection (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 1
Toxic shock syndrome streptococcal (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 2 | 0
Viral infection (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 0
Caustic injury (Injury, poisoning and procedural complications) | 1 | 0
Chest injury (Injury, poisoning and procedural complications) | 1 | 0
Compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 0
Device malfunction (Injury, poisoning and procedural complications) | 1 | 0
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 2 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Eye injury (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 8 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 | 0
Femur fracture (Injury, poisoning and procedural complications) | 4 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 8 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 0
Injury (Injury, poisoning and procedural complications) | 2 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 6 | 1
Joint dislocation postoperative (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 2 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Medical device complication (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Open fracture (Injury, poisoning and procedural complications) | 2 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 4 | 0
Radius fracture (Injury, poisoning and procedural complications) | 2 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 4 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 2 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 5 | 0
Wound (Injury, poisoning and procedural complications) | 2 | 0
Arteriogram coronary (Investigations) | 1 | 0
Blood pressure abnormal (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 1 | 0
Bone density decreased (Investigations) | 1 | 0
Cardiac ventriculogram left (Investigations) | 1 | 0
Catheterisation cardiac (Investigations) | 1 | 0
Heart rate abnormal (Investigations) | 1 | 0
Oxygen saturation decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 7 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Diabetic foot (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 4 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 2 | 0
Fracture delayed union (Musculoskeletal and connective tissue disorders) | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Hand deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Juvenile arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Low turnover osteopathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 15 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Pelvic deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 28 | 6
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 3 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 2 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 0
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 0
Colon cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Follicle centre lymphoma diffuse small cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gliosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Histiocytosis haematophagic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lentigo maligna stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0
Lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphocytic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to small intestine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prolymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain stem infarction (Nervous system disorders) | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Cerebral thrombosis (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 7 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 0
Hemiparesis (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 2 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0
Multiple sclerosis (Nervous system disorders) | 1 | 0
Radiculopathy (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 4 | 1
Transient ischaemic attack (Nervous system disorders) | 2 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Mental disorder (Psychiatric disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 3 | 0
Renal failure acute (Renal and urinary disorders) | 4 | 0
Renal tubular necrosis (Renal and urinary disorders) | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 0
Vaginal erythema (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diffuse alveolar damage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 2 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Panniculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 0
Joint prosthesis user (Social circumstances) | 1 | 0
Cardiac ablation (Surgical and medical procedures) | 1 | 0
Cholecystectomy (Surgical and medical procedures) | 1 | 0
Fracture treatment (Surgical and medical procedures) | 1 | 0
Hip arthroplasty (Surgical and medical procedures) | 1 | 0
Joint arthroplasty (Surgical and medical procedures) | 2 | 0
Knee arthroplasty (Surgical and medical procedures) | 4 | 0
Leg amputation (Surgical and medical procedures) | 1 | 0
Shoulder arthroplasty (Surgical and medical procedures) | 1 | 0
Shoulder operation (Surgical and medical procedures) | 1 | 0
Angiopathy (Vascular disorders) | 1 | 0
Aortic aneurysm rupture (Vascular disorders) | 2 | 0
Circulatory collapse (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 6 | 0
Haemorrhage (Vascular disorders) | 3 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 3 | 0
Infarction (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Peripheral embolism (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 0
Shock (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Total Adults (N=581) | Pediatric Subjects (N=58)
Abdominal pain (Gastrointestinal disorders) | 25 | 5
Abdominal pain upper (Gastrointestinal disorders) | 15 | 7
Diarrhoea (Gastrointestinal disorders) | 52 | 4
Dyspepsia (Gastrointestinal disorders) | 37 | 4
Nausea (Gastrointestinal disorders) | 40 | 5
Vomiting (Gastrointestinal disorders) | 13 | 4
Fatigue (General disorders) | 36 | 1
Injection site erythema (General disorders) | 65 | 8
Injection site pain (General disorders) | 3 | 3
Injection site pruritus (General disorders) | 39 | 3
Injection site swelling (General disorders) | 25 | 6
Pyrexia (General disorders) | 9 | 6
Bronchitis (Infections and infestations) | 89 | 4
Conjunctivitis infective (Infections and infestations) | 19 | 4
Cystitis (Infections and infestations) | 57 | 0
Ear infection (Infections and infestations) | 12 | 4
Gastroenteritis viral (Infections and infestations) | 17 | 4
Influenza (Infections and infestations) | 60 | 7
Otitis media (Infections and infestations) | 17 | 5
Pharyngitis (Infections and infestations) | 30 | 13
Pharyngitis streptococcal (Infections and infestations) | 5 | 5
Pneumonia (Infections and infestations) | 31 | 1
Sinusitis (Infections and infestations) | 121 | 8
Skin infection (Infections and infestations) | 84 | 9
Upper respiratory tract infection (Infections and infestations) | 207 | 36
Fall (Injury, poisoning and procedural complications) | 21 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 53 | 0
Dizziness (Nervous system disorders) | 36 | 3
Headache (Nervous system disorders) | 80 | 20
Migraine (Nervous system disorders) | 13 | 3
Insomnia (Psychiatric disorders) | 38 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 13 | 5
Rash (Skin and subcutaneous tissue disorders) | 50 | 7
Hypertension (Vascular disorders) | 35 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, the investigator agrees not to publish any results before the first multi-center publication.